CLINICAL TRIAL: NCT05735717
Title: Phase II, Open-Label, Prospective Study of T Cell Receptor Alpha/Beta Depletion (A/B TCD) Peripheral Blood Stem Cell (PBSC) Transplantation for Children and Adults With Hematological Malignancies
Brief Title: MT2021-08T Cell Receptor Alpha/Beta Depletion PBSC Transplantation for Heme Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS061
Record Dates: First submitted 2023-01-10; First posted 2023-02-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy; Acute Leukemia; Remission; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; AML; TP53; Intrachromosomal Amplification of Chromosome 21; Cytogenetic Abnormality; CNS Leukemia; Minimal Residual Disease; Myelodysplasia; Juvenile Myelomonocytic Leukemia; Somatic Mutation; PTPN11 Gene Mutation; N-RAS Gene Amplification; Neurofibromatosis 1; NF1 Mutation; CBL Gene Mutation; Monosomy 7; Chromosome Abnormality; Fetal Hemoglobin
Keywords: Bu; Flu; G-CSF; GFSR; aGVHD; HCT; MAC; Mel; PBSCT; PTLD; RECIST; TCR
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Chromosome Aberrations; Neoplasm, Residual; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Juvenile; Neurofibromatosis 1; Chromosome 7, monosomy; beta-Thalassemia; Influenza, Human | interventions — fludarabine; Busulfan; Melphalan; Rituximab; Levetiracetam; thymoglobulin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm 1A: Fludarabine (flu), Total Body Irradiation (TBI), Flu/TBI Regimen, Closed to Accrual (Experimental): Patients will be treated on the most medically appropriate regimen with a preference for Flu/TBI Arm followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Interventions: Drug: Fludarabine; Drug: Rituximab; Drug: Levetiracetam; Biological: Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells
- Arm 2A: Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen, Closed to Accrual (Experimental): Patients will be treated on the most medically appropriate regimen with a preference for Flu/TBI Arm followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Rituximab; Drug: Levetiracetam
- Arm 3A: Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only (Experimental): Flu/Bu/Mel will the preference for patients with JMML or infants with leukemia. , Closed to Accrual
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Melphalan; Drug: Rituximab; Drug: Levetiracetam
- Arm 1B: ATG, Fludarabine (flu), Total Body Irradiation (TBI), Flu/TBI Regimen (Experimental): Patients will be treated on the most medically appropriate regimen with a preference for ATG/Flu/TBI Arm followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Interventions: Drug: Fludarabine; Drug: Rituximab; Drug: Levetiracetam; Drug: Thymoglobulin
- Arm 2B: ATG, Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen (Experimental): Patients will be treated on the most medically appropriate regimen with a preference for ATG/Flu/BU/TBI Arm followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Rituximab; Drug: Levetiracetam; Drug: Thymoglobulin
- Arm 3B: ATG, Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only (Experimental): ATG/Flu/Bu/Mel will the preference for patients with JMML or infants with leukemia.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Melphalan; Drug: Rituximab; Drug: Levetiracetam; Drug: Thymoglobulin
- Arm 4B: ATG, Busulfan (BU), Cyclophosphamide (CY) (Experimental): Patients will be treated on the most medically appropriate regimen with a preference for ATG/BU/CY Arm followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Interventions: Drug: Busulfan; Drug: Rituximab; Drug: Levetiracetam; Drug: Thymoglobulin; Drug: Cyclophosphamide
- Arm 5B: ATG, Cyclophosphamide (CY), Total Body Irradiation (TBI) (Experimental): Patients will be treated on the most medically appropriate regimen with a preference for ATG/CY/TBI Arm followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Interventions: Drug: Rituximab; Drug: Levetiracetam; Drug: Thymoglobulin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 25mg/m2 IV on days -8 to -6 or days -4 to -2. 40mg/m2 IV on days -5 to -2.
  Arms: Arm 1A: Fludarabine (flu), Total Body Irradiation (TBI), Flu/TBI Regimen, Closed to Accrual; Arm 1B: ATG, Fludarabine (flu), Total Body Irradiation (TBI), Flu/TBI Regimen; Arm 2A: Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen, Closed to Accrual; Arm 2B: ATG, Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen; Arm 3A: Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only; Arm 3B: ATG, Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only
Drug: Busulfan — Busulfan 82.1 mg*hr/L IV on days -5 to -2 or days -8 to -5
  Arms: Arm 2A: Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen, Closed to Accrual; Arm 2B: ATG, Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen; Arm 3A: Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only; Arm 3B: ATG, Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only; Arm 4B: ATG, Busulfan (BU), Cyclophosphamide (CY)
Drug: Melphalan — Melphalan 50 mg/m2 IV on days -4 to -2
  Arms: Arm 3A: Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only; Arm 3B: ATG, Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only
Drug: Rituximab — 200 mg/m2 intravenous given once on day-1
Drug: Levetiracetam — As seizures have occurred following high dose busulfan, all patients will be treated with Keppra beginning day -6 and continuing until day -1 per institutional guidelines.
  Other Names: Keppra
Biological: Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells — Patients will be treated on the most medically appropriate regimen followed by an infusion at Day 0 of Alpha/Beta T Cell-Depleted Hematopoietic Stem Cells.
  Arms: Arm 1A: Fludarabine (flu), Total Body Irradiation (TBI), Flu/TBI Regimen, Closed to Accrual
Drug: Thymoglobulin — rabbit anti-thymocyte globulin (rATG). Used in conditioning regimens for in vivo depletion of T cells, and the use of fludarabine model-based dosing to optimize dosing.
  Other Names: ATG
  Arms: Arm 1B: ATG, Fludarabine (flu), Total Body Irradiation (TBI), Flu/TBI Regimen; Arm 2B: ATG, Fludarabine (flu), Busulfan (bu), Flu/Bu Regimen; Arm 3B: ATG, Fludarabine (flu), Busulfan (bu), Melphalan (Mel) Regimen for Pediatric Patients Only; Arm 4B: ATG, Busulfan (BU), Cyclophosphamide (CY); Arm 5B: ATG, Cyclophosphamide (CY), Total Body Irradiation (TBI)
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg IV over 2 hours on days -3 and -2
  Arms: Arm 4B: ATG, Busulfan (BU), Cyclophosphamide (CY); Arm 5B: ATG, Cyclophosphamide (CY), Total Body Irradiation (TBI)

SUMMARY:
This is a phase II, open-label, prospective study of T cell receptor alpha/beta depletion (TCR α/β TCD) peripheral blood stem cell (PBSC) transplantation for children and adults with hematological malignancies. This is a safety/feasibility study of the investigational procedure/product.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of hematological malignancies
* Acute leukemias
* Acute Myeloid Leukemia (AML) and related precursor neoplasms
* Favorable risk AML is defined as having one of the following:
* Acute lymphoblastic leukemia (ALL)/lymphoma
* Myelodysplasia (MDS) IPSS INT-2 or High Risk (i.e. RAEB, RAEBt) or Refractory Anemia with severe pancytopenia, transfusion dependence, or high risk cytogenetics or molecular features.
* Age 60 years of age or younger at the time of consent
* Karnofsky performance status ≥ 70% or Lansky play score 50% for ≤16 years of age.
* Adequate organ function

Exclusion Criteria:

* Pregnant or breastfeeding.
* Active uncontrolled infection within 1 week of starting preparative therapy
* Known seropositive for HIV or known active Hepatitis B or C infection with detectable viral load by PCR.
* Any prior autologous or allogeneic transplant
* CML blast crisis
* Active central nervous system malignancy

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of GVHD after alpha beta TCR depletion | 100 days
  GVHD incidence after treatment.

SECONDARY OUTCOMES:
Transplant engraftment | 42 days
  Monitor median rate of engraftment by 42 days.
Graft Failure | 100 days
  Determine the rate of graft failure by day 100 (defined as lack of achievement of an ANC >=500/mL with associated pancytopenia)
Non-relapse mortality (NRM) | 12 months
  Determine the incidence of non-relapse mortality (NRM) at 100 days and 1 year
Overall survival (OS) | 12 months
  Number of participants experiencing progression free survival at one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
For the purposes of data and safety monitoring, this study is classified as high risk (investigator initiated under an IND). Therefore the following requirements will be fulfilled:
  * The Masonic Cancer Center Data and Safety Monitoring Council (DSMC) will review the study's progress at least quarterly.
  * The PI will comply with at least twice yearly monitoring of the project by the Masonic Cancer Center monitoring services.
  * The PI will oversee the submission of all reportable adverse events per the definition of reportable in Section 11.5 to the Masonic Cancer Center's SAE Coordinator, the University of Minnesota IRB, and the FDA.